CLINICAL TRIAL: NCT00601432
Title: An Open-label, Randomized, 2-way Crossover Study to Evaluate the Effect of Food on Levofloxacin Pharmacokinetics From an Oral Solution Formulation
Brief Title: A Study to Evaluate the Effect of Food on Levofloxacin Pharmacokinetics From an Oral Solution Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR010621
Record Dates: First submitted 2007-12-06; First posted 2008-01-28 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: open-label; randomized; crossover; food effect
MeSH Terms: interventions — Levofloxacin

INTERVENTIONS:
Drug: levofloxacin oral solution

SUMMARY:
The main purpose of the study was to evaluate the effect of food on the single-dose pharmacokinetics of an oral solution of levofloxacin.

DETAILED DESCRIPTION:
In this single-dose study conducted at a single center, the effect of food on the pharmacokinetics of levofloxacin was studied in 24 healthy men and women aged 18 to 55 years old. Subjects were assigned different treatments based on chance; both the researcher and the study participant knew the treatment being administered. The study consisted of 3 phases: a screening phase, an open-label treatment phase consisting of 2 treatment periods, and a post-treatment phase. Subjects who met the prestudy eligibility criteria were randomly assigned to 1 of 2 treatment sequence groups. In each treatment period, subjects were admitted to the study facility the evening before study drug administration and housed through 48 hours after dosing with study drug. Subjects received levofloxacin as a single oral dose of 500 mg under both fed (within 10 minutes after completion of a high-fat, high-caloric breakfast) and fasted (10-hour overnight fast) conditions according to their randomized treatment sequence. Each dosing day was separated by a washout period of at least 4 days. In each treatment period, pharmacokinetic blood samples were collected immediately prior to dosing and at 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 10, 14, 24, 30, 36, and 48 hours after dosing for determination of plasma concentrations of levofloxacin. Safety evaluations, including adverse event monitoring, standard clinical laboratory evaluations (hematology, serum chemistry, and urinalysis), vital sign monitoring, and physical examinations were performed on Days 1 and 3 of each treatment period. The post-treatment phase consisted of safety evaluations performed after collection of the final pharmacokinetic blood sampling in the second treatment period. Adverse events were monitored from the time of the first study-related procedure through completion of post-treatment study procedures, or until the time of early withdrawal from the study. Levofloxacin solution administered as 2 single oral doses of 500 mg each, 1 in each treatment period, administered at least 4 days apart.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged 18 to 55 years
* BMI between 18 and 30 kg/m2
* No prescription or over-the-counter medication for previous 14 days
* Negative tests for drug and alcohol abuse
* HIV, hepatitis B and hepatitis C
* and Healthy based on medical history, physical examination, 12-lead electrocardiograms, toxicology, antigen, antibody screens, and clinical laboratory evaluations

Exclusion Criteria:

* Allergic reaction to quinolones
* clinically significant ECG or clinical laboratory abnormalities
* creatinine clearance <=80 mL/min
* acute illness within 7 days
* receipt of experimental drug or device within 60 days
* pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-10; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of food on the single-dose pharmacokinetics of an oral solution of levofloxacin at 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 10, 14, 24, 30, 36, and 48 hours after dosing.

SECONDARY OUTCOMES:
Safety was assessed through vital sign monitoring, physicals, laboratory tests, and urinalysis on Days 1 and 3 and through the monitoring of adverse events throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An open-label, randomized, 2-way crossover study to evaluate the effect of food on levofloxacin pharmacokinetics from an oral solution formulation — http://download.veritasmedicine.com/PDF/CR010621_CSR.pdf